CLINICAL TRIAL: NCT00338494
Title: Dose Escalation Study of Clofarabine in Patients With Relapsed or Refractory Low Grade or Intermed.Grade B-Cell/T-Cell Lymphoma
Brief Title: Dose Escalation Study of Clofarabine in Patients With Relapsed or Refractory Low Grade or Intermediate-Grade B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0506000158
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — The starting dose of clofarabine will be 10 mg/m2 once a week for 3 weeks repeated every 4 weeks with dose escalations to 15, 20 , 30 and 40 mg/m2/week.
  Other Names: CAFdA; Cl-F-ara-A

SUMMARY:
Clofarabine is a new chemotherapy drug which was FDA approved for the treatment of acute lymphocytic leukemia in children. This study is being done to see if Clofarabine works in adult patients with B-cell types of lymphoma.

This research is being done to develop new treatments for patients with lymphoma whose cancer has returned or resisted treatment with previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are at least 18 years old
* Histologically confirmed low grade or intermediate-grade B-cell lymphoma
* Relapsed or refractory to at least one standard chemotherapy regimen. Patients who have received Rituximab alone without having received a cytotoxic agent are not eligible.
* Measurable disease, defined by the Cheson lymphoma criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy greater than 12 weeks
* Laboratory values obtained ≤2 weeks prior to entry

  * Absolute neutrophil count (ANC) ≥ 1000 x 10 9/L
  * White blood cell (WBC) count > 2.5 x 10 9/L
  * Platelets ≥ 75 x 10 9/L
  * Hemoglobin (Hg) > 9.0 g/dL
  * Total bilirubin ≤2.0 mg/dL
  * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤3 × upper limit of normal (ULN)
  * Serum creatinine ≤2.0 mg/dL
* Normal cardiac function, defined as an ejection fraction ≥45% determined by pretreatment radionuclide ventriculography (RVG) or echocardiogram.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Previously untreated B-cell lymphoma.
* Received previous treatment with clofarabine.
* Patients with known AIDS-related or HIV-positive lymphoma.
* Autologous bone marrow or stem cell transplant within 6 months of study entry.
* Prior radiotherapy to the only site of measurable disease.
* Any medical condition that requires chronic use of oral high-dose corticosteroids greater than 20 mg/day prednisone.
* Active autoimmune thrombocytopenia.
* Use of investigational agents within 30 days or any anticancer therapy within 3 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy.
* Patients with an active, uncontrolled systemic infection considered to be opportunistic, life threatening, or clinically significant at the time of treatment or with a known or suspected fungal infection (ie, patients on parenteral antifungal therapy).
* Active secondary malignancy.
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with active or untreated central nervous system (CNS) lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-10; Primary Completion 2010-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
tolerated dose (MTD) of clofarabine | at the completion of dose escalation
characterize and quantify the toxicity profile associated with clofarabine | upon completion of the study
determine the overall response rate, plus partial response of clofarabine | upon completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States